CLINICAL TRIAL: NCT02619149
Title: Piperacllin Versus Placebo in Patients Undergoing Surgery for Acute Cholecystitis
Acronym: AVAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AVAC
Record Dates: First submitted 2015-11-26; First posted 2015-12-02 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Piperacillin, Tazobactam Drug Combination; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Piperacillin-tazobactam combination product
  Interventions: Drug: Piperacillin-tazobactam combination product
- Control (Placebo Comparator): Saline solution
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Piperacillin-tazobactam combination product — Piperacillin-Tazobactam (extended-spectrum, beta-lactamase inhibitor) iv peroperatively as prophylaxis
  Other Names: Piperacillin-Tazobactam
  Arms: Intervention
Drug: Saline solution — Saline iv as placebo control
  Arms: Control

SUMMARY:
The benefit from antibiotic prophylaxis in patients undergoing laparoscopic cholecystectomy for acute cholecystitis is insufficiently known. The aim of the present double-blind randomized controlled is to compare piperacilin with placebo in patients undergoing cholecystectomy for acute cholecystitis with anamnesis not exceeding 5 days. Altogether 100 patients are intended to be included. Primary endpoint is biliary contamination. Secondary endpoints are postoperative hospital stay, health-related quality of life, pain perception, postoperative markers of inflammatory response, surgical site infections, infectious complications other than surgical site infections, health economy and relationship between symptom anamnesis and bile contamination.

DETAILED DESCRIPTION:
Background

Inflammation in the gallbladder due to obstruction of gallstones (acute cholecystitis) is a common condition and one of the most common indications for laparoscopic cholecystectomy. In most cases, the procedure may be performed without great risk of severe complications. In some cases, however, the congested bile in the gallbladder may become infected.

In clinical routine, acute cholecystitis is often managed as an infectious condition, despite the fact that previous studies have shown that the bile in most cases of acute cholecystitis is sterile. On the other hand, antibiotic prophylaxis may reduce the risk of surgical site infections in those cases when there is a manifest bacterial contamination and, perhaps, also reduce the risk of contamination. There is firm evidence supporting acute surgery, prefereably laparoscopic cholecystectomy, but the benefit from antibiotic treatment has not been full evaluated.

Previous studies have shown that the benefit from antibiotic prophylaxis is very limited in case of laparoscopic cholecystectomy for uncomplicated gallstone disease. There are, however, very few studies that have assessed antibiotic prophylaxis in surgery for acute cholecystitis.

The aim of the present study is to assess the benefit of antibiotic prophylaxis in patients undergoing laparoscopic cholecystectomy for acute cholecystitis.

Methods The study is based on patients admitted for acute cholecystitis at the department of acute surgery, Karolinska University Hospital Huddinge. In case the patients fulfill the inclusion critera and are suitable for laparoscopic surgery, written and oral information about the study is given.

In case they agree to participate in the study, treatment allocation is determined by a sealed envelope system. The patients are randomised to receive either Piperacillin 4g x 3 iv preoperatively as prophylaxis or placebo (saline infusion). The study is double-blind. Piperacillin/placebo is administrated by a research nurse after allocation. The infusion is covered by a bag in order to maintain blinding. Neither the surgeon performing the procedure, nor the patient or staff caring for the patient are informed about the allocation. The procedure should be performed within 24 days after inclusion. Administration of Piperacillin/placebo is started immediately after inclusion and continued until the procedure is completed.

If a categorical indication for antibiotic treatment occurs during surgery, the allocated infusion is removed and the patient is given antibiotic as decided by the surgeon. In such cases, the patient stays in the study and is analysed according to an intention to treat.

During the laparoscopic cholecystectomy, at least 10 cc of bile is aspirated under sterile conditions from the fundus of the gallbladder with a long needle before the start of the peritoneum dissection. The bile is sent for aerobic and anaerobic culture. Bacteria are identified using standard laboratory procedures.

Sample size estimation If the incidence of positive cultures is 50% and in the placebo group and this is reduced to 25% if antibiotic prophylaxis is given, 36 patients in each arm would be required in order to reach 80% chance of detecting this difference at a p<0.05 level of significance (one sided test). A total sample of 100 patients should thus be sufficient to test the primary outcome measure.

Follow-up Samples for CRP, interleukins, bilirubin, AST, ALT and ALP are taken daily from the peroperative day until postoperative day 2.

Quality of life is assessed by SF-36 preoperatively. Level of pain is estimated based on the MacGill Pain Questionnaire from the day of the procedure until postoperative day 2.

One month postoperatively, the patient is invited to follow-up. At follow-up, SF-36 is filled in.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiologic signs of acute cholecystitis
* First acute symptoms occurring within five days before surgery

Exclusion Criteria:

* Anamnesis exceeding five days
* Any contraindication for laparoscopic surgery
* Allergy against beta-lactame antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Proportion of positive bacterial cultures | 5 days
  Proportion of patients with bacterial growth in the bile, assessed by culture from the bile assembled perioperatively.

SECONDARY OUTCOMES:
Postoperative hospital stay | 5-10 days
Health-related quality of life | One month
  Health-related quality of Life measured with SF-3
Postoperative pain as measured by the McGill Pain Questionnaire | 3 days
  Level of pain as measured by the McGill Pain Questionnaire
Levels of C-reactive Protein postoperatively | 3 days
  CRP levels measured daily in the postoperative period
Surgical site infections | 5-10 days
  Abscesses or superficial wound infections requiring drainage or antibiotic treatment
Infectious complications other than surgical site infections | 5-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Folke Hammarqvist, Ass Prof, Principal Investigator — Karolinska Institutet, CLINTEC, Stockholm
Locations (1):
- Karolinska University Hospital, Center for Digestive Diseases, Stockholm, Sweden

REFERENCES:
- [Derived] Jaafar G, Sandblom G, Lundell L, Hammarqvist F. Antibiotic prophylaxis in acute cholecystectomy revisited: results of a double-blind randomised controlled trial. Langenbecks Arch Surg. 2020 Dec;405(8):1201-1207. doi: 10.1007/s00423-020-01977-x. Epub 2020 Aug 29. PMID 32860109